CLINICAL TRIAL: NCT00165503
Title: A Phase II Feasibility Study of Pleurectomy/Decortication With Intraoperative Intrathoracic/Intraperitoneal Heated Cisplatin With Sodium Thiosulfate Followed ny Adjuvant ALIMTA/Cisplatin
Brief Title: Pleurectomy/Decortication With Intraoperative Intrathoracic/Intraperitoneal Heated Cisplatin With Sodium Thiosulfate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of acurral
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David J. Sugarbaker, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-063
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-07

CONDITIONS: Pleural Mesothelioma; Malignant Pleural Mesothelioma
Keywords: pleurectomy; decortication; cisplatin; ALIMTA
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; sodium thiosulfate; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery+Heated Cisplatin+Sodium Thiosulfate+Adjuvant CT (Experimental): Participants undergo surgery, Pleurectomy/Decortication, followed by heated cisplatin given as a one-hour lavage of the chest and abdominal cavity then sodium thiosulfate given intravenously over 6 hours. The adjuvant chemotherapy regimen beginning 6-10 weeks after surgery is a combination of cisplatin and Alimta each given day 1 of a 21-day cycle for 3 cycles.
  Interventions: Drug: Cisplatin; Drug: Sodium Thiosulfate; Drug: ALIMTA

INTERVENTIONS:
Drug: Cisplatin
Drug: Sodium Thiosulfate
Drug: ALIMTA
  Other Names: pemetrexed

SUMMARY:
The purposes of this study are: to determine the feasibility of administering adjuvant cisplatin plus ALIMTA to patients who undergo surgery with heated cisplatin during surgery; to determine the effects (good and bad) of this combined modality approach in patients with mesothelioma; to evaluate cisplatin effects by determining where it goes and how it is excreted in the body from the collection of tissues and cisplatin samples; to collect and analyze discarded samples of mesothelioma tumor during surgery to help determine the genetic make-up of the disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of administering adjuvant cisplatin plus Alimta to patients undergoing surgery with hyperthermic cisplatin.

Secondary

* To determine the morbidity and mortality of this treatment protocol
* To determine time to tumor recurrence and patient survival
* To evaluate the pharmacokinetics of intraoperatively administered cisplatin

DETAILS:

* Patients will undergo surgery, which is part of the standard care for mesothelioma, by a procedure called pleurectomy/decortication. This involves removal of the lining of the lung and all visible disease. Resection of the lining of the heart and the muscle that separates the chest and abdomen is occasionally necessary.
* Mesothelioma samples will be taken during the surgery. These samples will be used in a laboratory study to better understand the genetic makeup of the mesothelioma and to improve our ability to diagnose this disease.
* After the conclusion of the surgery, if a patient has less than 1cm thickness of residual gross disease in one or more areas, then the patient will continue on this study. If more than this volume of tumor is present, then the patient will receive additional treatment off-study.
* Heated chemotherapy (cisplatin) will be given in the operating room immediately following surgery. This treatment consists of a one-hour lavage of the chest and abdominal cavity with heated cisplatin through the surgical incision. At the completion of the hour, sodium thiosulfate is given intravenously for 6 hours to reduce potential side effects.
* During the surgery and for four hours following the completion of the cisplatin lavage, blood samples, urine samples, chest wall muscle samples, and samples of the chemotherapy solution will be taken in order to measure the concentration of chemotherapy and the impact of cisplatin in these samples.
* Patients will remain in the hospital until they have recovered from surgery (7-14 days). In addition to standard post-operative care, blood tests will be done on a daily basis. Following discharge from the hospital, patients will be seen 1-2 weeks post-operatively for additional blood work. An echocardiogram will be done 6 weeks and 6 months post-operatively to assess heart function.
* Chemotherapy treatment consists of ALIMTA plus cisplatin on Day 1 of every 21-day chemotherapy cycle. A total of 3 cycles will be given starting 6-10 weeks after surgery.
* Folic acid, vitamin B12 and dexamethasone will be given in addition to the chemotherapy to help reduce side effects of the chemotherapy drugs.
* Approximately 30 days after the last dose of ALIMTA plus cisplatin, a CT scan(s) and blood work will be performed. In addition, patients will get a CT scan(s) every 3 months for approximately 24 months from the completion of study treatment.
* Long term follow-up will consist of clinic visits every 3 months for 2 years, every 6 months for 2 years, and then once a year.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic confirmation of malignant pleural mesothelioma
* Patients who are able to tolerate surgical cytoreduction but unable to undergo extrapleural pneumonectomy due to poor cardiopulmonary reserve or tumor invasion or those with minimal disease
* Male on non-pregnant female
* 18 years of age or older
* No evidence of spread outside the ipsilateral hemithorax by chest CT and chest MRI
* Ejection fraction > 45%
* Pre-operative WBC > 4K/uL
* Estimated life expectancy of at least 12 weeks
* Evidence of adequate renal and hepatic function
* Grossly normal contralateral pulmonary function with a chest radiograph and chest CT scan
* Karnofsky performance status of 70% or greater
* No evidence of disease progression by chest CT or chest MRI, obtained at 8 weeks following surgery

Exclusion Criteria:

* Extended disease outside the ipsilateral hemithorax as determined on pre-operative radiographs or intraoperative findings
* Positive extrapleural nodes as determined by mediastinoscopy
* Gross disease (estimated thickness > 10mm at any intrathoracic location) present within the hemithorax after surgery
* Evidence of distant metastatic disease
* Severe non-malignant co-morbid disease, uncontrolled angina, myocardial infarction on the past 6 months, renal insufficiency, liver disease, pulmonary hypertension
* Pregnant or breast-feeding
* Serious concomitant systemic disorders
* Presence of active concomitant malignancy
* Psychiatric or addictive disorders, which would preclude informed consent
* Previous chemotherapy or radiation therapy for mesothelioma
* Chemotherapy or radiation therapy administered within 3 years for another malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Sugarbaker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin, Sodium Thiosulfate, Alimta: Heated Cisplatin will be given as a one-hour lavage of the chest and abdominal cavity following surgery.Cisplatin will also be administered intravenously as part of chemotherapy 6-10 weeks after surgery. It will be given on day 1 of each 21-day treatment cycle for 3 cycles. Sodium Thiosulfate Given intravenously over 6 hours following heated cisplatin lavage. Alimta Given intravenously on day 1 of each 21-day treatment cycle for a total of 3 cycles beginning 6-10 weeks after surgery.
Period: Overall Study
Arm/Group | Cisplatin, Sodium Thiosulfate, Alimta
Started | 16
Completed | 0
Not Completed | 16
Not completed — Death | 1
Not completed — Lost to Follow-up | 12
Not completed — Unresectable | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin, Sodium Thiosulfate, Alimta
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 71.5 [45 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0
  Non-Hispanic | 16
Region of Enrollment [Number; unit: participants]
  United States | 15
  Israel | 1

OUTCOME MEASURES:

1. Primary Outcome: Adjuvant Chemotherapy Completion Rate
Description: Feasibility in this study was based on the adjuvant chemotherapy regimen. The chemotherapy completion rate is defined as the percentage of patients who complete 3 cycles of cisplatin and Alimta beginning 6-10 weeks after surgery with hyperthermic cisplatin.
Time Frame: Given the 21-day cycle, 3 cycles of adjuvant chemotherapy approximates 9 weeks in addition to the time from registration and post-surgery which was up to 10 weeks.
Population: None of the enrolled participants were evaluated for the primary endpoint since none received the experimental adjuvant chemotherapy per protocol.
Arm/Group | Surgery+Heated Cisplatin+Sodium Thiosulfate+Adjuvant CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The period for reporting adverse events were 30 days from the participant's date of surgery.
Groups:
- Surgery + Heated Cisplatin Lavage + Sodium Thiosulfate: Participants undergo surgery, Pleurectomy/Decortication, followed by heated cisplatin given as a one-hour lavage of the chest and abdominal cavity then sodium thiosulfate given intravenously over 6 hours.
Arm/Group | Surgery + Heated Cisplatin Lavage + Sodium Thiosulfate
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgery + Heated Cisplatin Lavage + Sodium Thiosulfate (N=16)
Pericardial effusion with tamponade (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Progression of disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypocalcemia (Blood and lymphatic system disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Elevated troponin (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
This trial was terminated due to low accrual and feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes